CLINICAL TRIAL: NCT05328622
Title: Rewarding Healthy Behaviors in Pregnancy and Postpartum With Aqueduct
Brief Title: Rewarding Healthy Behaviors in Pregnancy and Postpartum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Transcendent International, LLC (Industry)
Collaborators: MOUNT SINAI HOSPITAL (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HHS-1R44NR020320-01A1
Record Dates: First submitted 2022-03-24; First posted 2022-04-14 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Pregnancy Related
Keywords: Postpartum; Adherence; Prenatal

STUDY DESIGN:
Intervention Model Description: All participants will receive daily text messages and incentives for medical adherence. Recruitment will occur on a rolling basis, with participants completing the protocol in multiple waves.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adherence Incentives Program (Experimental): The intervention administered to participants is an incentive program designed to motivate participants to attend to/adhere to their prescribed prenatal course of care via the Aqueduct platform.
  Interventions: Behavioral: Aqueduct Contingency Management Platform

INTERVENTIONS:
Behavioral: Aqueduct Contingency Management Platform — All individuals who consent to participate will engage with the Aqueduct contingency management system. Once participants are enrolled, they accumulate points in Aqueduct for each prenatal/postpartum appointment they attend. They also earn points for attending pregnancy and birth related classes, monitoring their health (e.g., blood sugar, blood pressure), and taking prescribed medications. Participants then redeem their points for money on a Visa gift card.
  Enrolled participants also receive daily text messages that contain motivational and mini-educational content regarding pregnancy from trusted sources such as the American College of Obstetricians and Gynecologists, Evidence Based Birth, and Postpartum Support International. These texts serve as reminders to participants to remain engaged in their pregnancy care.

SUMMARY:
This is a single-arm pilot clinical trial with two primary research goals:

1. To test the efficacy of a software's ability to profile eligible individuals who decline participation in a clinical trial ("non-consenters") so that research staff may improve recruitment strategies for subsequent waves of potential participants.
2. To test the feasibility of using the software's contingency management program in a population of pregnant persons in their third trimester of pregnancy.

DETAILED DESCRIPTION:
The first aim of the study is to test the feasibility of using a software program to incentivize pregnant patients to adhere to their prescribed prenatal appointments, postnatal appointment, and healthy behaviors. Participants will receive daily text messages that encourage engagement with health behaviors, and then participants earn points when they attend their scheduled appointments, bring in prescribed monitoring logs, and take their medications as prescribed.

A related aim of the study is to examine the effectiveness of the software system in providing support to researchers in implementing targeted participant recruitment in a manner that is labor-efficient and sustainable. The study will determine the efficacy of the software for (1) using psycho-demographic data to achieve more representative enrollment vis-à-vis target populations and (2) iteratively tailoring outreach materials and communication techniques based on actionable insights about those who participate and those who decline to participate.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant in third trimester of pregnancy
* Between 18 and 52 years of age
* Able to read and speak either English or Spanish
* A patient at Mount Sinai Hospital's OB-Gyn Ambulatory E-Level Clinic

Exclusion Criteria:

* Not pregnant (or no longer pregnant)
* Outside of age range
* Unwilling or unable to complete surveys
* Not a patient at the clinic of interest

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Percentage of prenatal appointments attended | 4 months
  Using data from Mt. Sinai's electronic medical record appointment tracking system, the investigators will determine whether participants who received the Aqueduct system intervention demonstrate increased attendance at scheduled prenatal visits compared with baseline data in the clinic about attendance rates.
Percentage of postpartum appointments attended | 4 months
  Using data from Mt. Sinai's electronic medical record appointment tracking system, the investigators will determine whether participants who received the Aqueduct system intervention demonstrate increased attendance at scheduled postpartum visits compared with baseline data in the clinic about attendance rates.
Percentage of eligible target population who consent to participate | 4 months
  Using descriptive statistics from recruitment, the investigators will determine whether the percentage (%) of eligible individuals from the population of pregnant women in their third trimester receiving prenatal care at the Mt. Sinai E-Level OB Clinic who elected to participate in the study increases between Wave 1 and Wave 2 of recruitment based upon changes in recruitment language.

SECONDARY OUTCOMES:
Changes in healthy eating between baseline and follow-up | 4 months
  Using self-reported frequency of eating fruits, vegetables, and fried foods (measured as average number of days per week over the past month), the investigators will determine whether participants who received the Aqueduct system intervention demonstrate increased frequency in consumption of fruits and vegetables, as well as decreased fried food consumption, from baseline (start of third trimester) to follow-up (postpartum appointment ~6 weeks after giving birth).
Changes in exercise habits between baseline and follow-up | 4 months
  Using self-reported number of minutes of moderate intensity physical activity (measured as average minutes per week over the past month), the investigators will determine whether participants who received the Aqueduct system intervention demonstrate increased minutes of physical activity from baseline (start of third trimester) to follow-up (postpartum appointment ~6 weeks after giving birth).
Changes in self-efficacy between baseline and follow-up | 4 months
  Using the General Self-Efficacy questionnaire, the investigators will determine whether participants who received the Aqueduct system intervention demonstrate increased self-efficacy from baseline (start of third trimester) to follow-up (postpartum appointment ~6 weeks after giving birth). Respondents use a 5-point rating scale (1= strongly disagree; 3 = neither agree nor disagree; 5 = strongly agree). Total scores range from 8 - 40, with higher total scores indicating better/stronger self-efficacy. Instrument citation: Chen, G., Gully, S. M., & Eden, D. (2001). Validation of a new general self-efficacy scale. Organizational Research Methods, 4(1), 62-83. Accessed via https://sparqtools.org/mobility-measure/new-general-self-efficacy-scale/#all-survey-questions

CONTACTS AND LOCATIONS:
Overall Officials: Aviva H Ariel-Donges, PhD, MPH, Study Director — Transcendent Endeavors
Locations (1):
- Mount Sinai Hospital OB-Gyn Clinic E-Level, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No